CLINICAL TRIAL: NCT03189732
Title: New Electrophoretic Approaches in Studies of Obesity and Diabetes
Brief Title: Effect of Metformin on Exercise-induced Lipolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Vladimir Stich, Professor, MUDr, Charles University, Czech Republic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15-03139S
Record Dates: First submitted 2017-05-31; First posted 2017-06-16 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: lipolysis; adipose tissue; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Metformin; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metformin oral +exercise (Experimental): Metformin, one dose 2000mg, 2.5h before the start of 60 min physical exercise
  Interventions: Drug: Metformin Oral; Other: Exercise
- Metformin local in AT +exercise (Active Comparator): Metformin perfused into microdialysis probe inserted in adipose tissue, 0.3ug/min 1.5h before the exercise and during 60min physical exercise
  Interventions: Drug: Metformin local in AT; Other: Exercise
- No metformin + exercise (Active Comparator): 60min physical exercise without pretreatment of metformin
  Interventions: Other: Exercise

INTERVENTIONS:
Drug: Metformin Oral
  Other Names: Metformin tablet
  Arms: Metformin oral +exercise
Drug: Metformin local in AT
  Other Names: Metformin dialysate
  Arms: Metformin local in AT +exercise
Other: Exercise
  Other Names: Acute exercise

SUMMARY:
The aim of this study is to investigate whether metformin has inhibitory effect on exercise-induced lipolysis in subcutaneous adipose tissue in healthy lean man. Ten healthy lean mean will follow protocols consisting of 60 minutes of exercise on bicycle ergometer combined with a) orally administered metformin and b) locally administered metformin into adipose tissue and c) without metformin treatment. Microdialysis is used for assessment of metabolites in situ in subcutaneous adipose tissue.

DETAILED DESCRIPTION:
Metformin and physical activity are often recommended as the first therapeutic agents to improve glycemic control for prediabetes and type 2 diabetes (ADA). It has been reported that metformin decrease plasma concentration of non-esterified fatty acids in patients with type 2 diabetes which might be associated with the inhibition of lipolysis in adipose tissue. However, the inhibition of lipolysis during physical exercise, would not be probably beneficial. Thus, the effect of metformin on lipolysis during exercise is investigated in this protocol. As the lipolysis regulation is often impaired in obese and diabetic patients, the healthy lean men were chosen for this pilot study. Glycerol will be analyzed as a measure of lipolytic rate in adipose tissue and in plasma. Lactate levels will be observed. Our findings should provide a new background about the combination of physical activity and metformin medication.

ELIGIBILITY:
Inclusion Criteria:

* healthy lean men, non obese, BMI 20-28 kg/m2

Exclusion Criteria:

* weight change within the 3 months before the study,
* hypertension,
* impaired fasting glucose
* diabetes
* hyperlipidemia
* drug or alcohol abuse
* smoking

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in adipose tissue lipolysis in response to exercise | Minute -60, 15, 30, 45, 60 and 120 from the start of exercise
  Glycerol concentration in dialysate outcoming from adipose tissue and in plasma - kinetic study

SECONDARY OUTCOMES:
Change in lactate production in response to exercise | Minute -60, 15, 30, 45, 60 and 120 from the start of exercise
  Concentration of lactate in dialysate and in plasma - kinetic study

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Stich, prof, Study Chair — Third faculty of medicine, Charles University in Prague
Locations (1):
- Third Faculty of Medicine, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bourron O, Daval M, Hainault I, Hajduch E, Servant JM, Gautier JF, Ferre P, Foufelle F. Biguanides and thiazolidinediones inhibit stimulated lipolysis in human adipocytes through activation of AMP-activated protein kinase. Diabetologia. 2010 Apr;53(4):768-78. doi: 10.1007/s00125-009-1639-6. Epub 2009 Dec 31. PMID 20043143
- [Background] Flechtner-Mors M, Ditschuneit HH, Jenkinson CP, Alt A, Adler G. Metformin inhibits catecholamine-stimulated lipolysis in obese, hyperinsulinemic, hypertensive subjects in subcutaneous adipose tissue: an in situ microdialysis study. Diabet Med. 1999 Dec;16(12):1000-6. doi: 10.1046/j.1464-5491.1999.00189.x. PMID 10656228
- [Background] Ren T, He J, Jiang H, Zu L, Pu S, Guo X, Xu G. Metformin reduces lipolysis in primary rat adipocytes stimulated by tumor necrosis factor-alpha or isoproterenol. J Mol Endocrinol. 2006 Aug;37(1):175-83. doi: 10.1677/jme.1.02061. PMID 16901933